CLINICAL TRIAL: NCT01117129
Title: Efficacy of MabThera in Patients With Rheumatoid Arthritis, by Measurement of Disease Parameters Through Magnetic Resonance of the Hand (RESONAR Study)
Brief Title: A Study of Efficacy of Rituximab [Mabthera/Rituxan] in Patients With Rheumatoid Arthritis Using Magnetic Resonance Imaging of the Hand (RESONAR)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was prematurely terminated as 2 patients were recruited and both of them withdrawn from the study before reaching the primary end point.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ML21826; 2008-002381-55
Record Dates: First submitted 2010-05-04; First posted 2010-05-05 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]; Drug: methotrexate
- B (Placebo Comparator)
  Interventions: Drug: placebo; Drug: methotrexate; Drug: rituximab [Mabthera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000 mg by i.v. infusion on day 1 and 15
  Arms: A
Drug: placebo — i.v. infusion on day 1 and 15
  Arms: B
Drug: methotrexate — 10-25 mg weekly
Drug: rituximab [Mabthera/Rituxan] — 1000 mg by i.v. infusion on day 1 and 15, 2nd and further cycles in patients with (group A) or without (group B) clinical response in cycle 1

SUMMARY:
This randomized, double-blind, placebo controlled, parallel group study will assess the efficacy and safety of rituximab [MabThera/Rituxan] in patients with severe active rheumatoid arthritis refractory to at least one anti-TNF treatment, using magnetic resonance imaging (MRI) of the hand for efficacy measurement. Patients will be randomized to receive 2 intravenous infusions 14 days apart of either 1000mg MabThera (group A) or placebo (group B). All patients will receive methotrexate 10-25mg weekly. Patients in group A demonstrating clinical response at week 24 may receive further cycles of MabThera, patients in group B without clinical response will also be treated with active MabThera. Anticipated time on study treatment is up to 2 years. Target sample size is <50 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age
* active rheumatoid arthritis (DAS28-CRP>3.2)
* refractory to one or more anti-TNF
* on stable treatment for RA for >/=4 weeks
* evidence of erosive disease and/or synovitis in wrist and/or knuckles

Exclusion Criteria:

* active systemic or local infection
* previous or current history of any demyelinization process in central nervous system, pancytopenia or aplasic anaemia
* signs of immunodeficiency, HIV infection or tuberculosis
* contraindications to MRI, such as metal devices, claustrophobia, moderate or severe renal insufficiency, or allergy to contrast agent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Bone erosion score on magnetic resonance imaging (MRI) using the rheumatoid arthritis magnetic resonance imaging scoring system (RAMRIS) | 6 months

SECONDARY OUTCOMES:
Synovitis score on MRI using RAMRIS | months 6, 12 and 24
Bone edema score on MRI using RAMRIS | months 6, 12 and 24
Bone erosion score on MRI using RAMRIS | months 12 and 24
Disease activity according to DAS28-CRP | months 12 and 24
Tender or swollen joint count (ACR criteria) | months 12 and 24
Health assessment questionnaire (HAQ) | months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Barcelona, Barcelona, Spain